CLINICAL TRIAL: NCT07086339
Title: A Two Center Trial of the Implantable Artificial Bronchus 50 Flex (IAB 50 Flex) in Patients With Severe Emphysema
Brief Title: A Trial of the Implantable Artificial Bronchus 50 Flex in Patients With Severe Emphysema
Acronym: IAB-3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmair Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAB3-CIP-v01
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: COPD; Emphysema
Keywords: IAB; Pulmair Medical; Emphysema; COPD; Lung Volume Reduction; Interventional Pulmonology; Pulmonology; COPD treatment; Emphysema treatment; lung conditions; Lung disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): One or two procedures involving placement of up to 10 IAB implants in one or both lungs
  Interventions: Device: Implantable pulmonary stent

INTERVENTIONS:
Device: Implantable pulmonary stent — Implantable polymer based pulmonary stent for severe COPD/emphysema

SUMMARY:
A Study at Two Hospitals Testing the Safety and Effectiveness of the IAB 50 Flex, a New Implant for Adults with Severe COPD or Emphysema

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Diagnosis of COPD/emphysema
3. At least 22-years of age
4. 18 ≤ BMI ≤ 32
5. 6-minute walk Distance of between 100 - and 400 meters
6. Stable disease with less than 10-mg prednisone (or equivalent) daily
7. Non-smoking for 4-months prior to screening interview (this includes tobacco, vaping, marijuana, etc.).
8. FEV1 between 15% and 45% of predicted value at baseline exam
9. FEV1/FVC <70%
10. Subject has ≥25% emphysema destruction score in each lung defined by areas of low attenuation less than -950 HU, as determined by CT core lab.
11. Subject has homogeneous or heterogeneous emphysema, and at least one lung has a 15% difference between upper and lower lobes in emphysema destruction score less than -950 HU, as determined by CT core lab.
12. RV > 175% of predicted value.
13. mMRC score ≥ 2

Exclusion Criteria:

1. Currently participating in another clinical study that involves surgery, interventional or pharmaceutical treatment
2. α-1 Antitrypsin deficiency
3. Women of child-bearing potential
4. More than 2 COPD exacerbation episodes requiring hospitalization in the last year prior to screening
5. Any COPD exacerbations requiring hospitalization within 6-weeks of planned intervention
6. Two or more instances of pneumonia episodes requiring hospitalization in the last year prior to screening
7. Clinically significant mucus production or chronic bronchitis
8. Myocardial Infarction or unstable / uncontrolled congestive heart failure within 6-months of screening
9. Prior lung transplant, LVRS, bullectomy, lobectomy or endoscopic lung volume reduction (ELVR)
10. Clinically significant bronchiectasis
11. Unable to safely discontinue anti-coagulants or platelet activity inhibitors for 7-days
12. Uncontrolled pulmonary hypertension (systolic pulmonary arterial pressure >45 mm Hg) or evidence or history of cor pulmonale as determined by recent echocardiogram
13. Suspected malignant pulmonary nodule or other lung cancer
14. HRCT collected per CT scanning protocol within the last 6 months of screening date and evaluated by clinical site personnel using 3D segmentation software shows:

    * Large bullae encompassing greater than 30% of either lung
    * Insufficient landmarks to evaluate the CT study using the software as it is intended
    * All lobes are less than 25% parenchyma diseased (< -950 HU).
15. Any cardiac comorbidity which the PI believes would compromise the safety of the patient after an IAB implant
16. TLC < 100% predicted at screening
17. DLCO < 15% or > 50% of predicted value at screening
18. PaCO2 > 50 mm Hg at screening
19. PaO2 < 45 mm Hg in room air at screening
20. Plasma cotinine level > 13.7 ng/ml or carboxyhemoglobin (arterial or ear lobe capillary) >2.5% at screening.
21. Current diagnosis of substance abuse disorder.
22. Current diagnosis of any of the following: Major Depressive Disorder (MDD), Schizoaffective Disorder, Schizophrenia, Borderline Personality Disorder, Bipolar Disorder
23. Any other conditions, which, in the opinion of the Investigator, would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events | Ninety (90) days from the last IAB implanted.
  The incidence of respiratory serious adverse events related to the device or procedure (SADEs) through the 90-day endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No